CLINICAL TRIAL: NCT02956369
Title: Chronic Effect of Daily Intake of SATIOSTAT Over 6 Weeks on Weight Loss, Glucose Tolerance, Gastrointestinal Tolerance and Gut Microbiota.
Brief Title: Effect of Daily Intake of SATIOSTAT Over 6 Weeks on Weight Loss, Glucose Tolerance, Gastrointestinal Tolerance and Gut Microbiota.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SATIOSTAT chronic effects
Record Dates: First submitted 2016-11-02; First posted 2016-11-07 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — CD36 Antigens; Carbohydrates; Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): 10 obese, non-diabetic candidates will serve as control-group. All assessments are carried out just as in the intervention groups. The control granulates consists of maize starch and long-chain fatty acids with powder.
  Interventions: Dietary Supplement: Control
- SATIOSTAT (Active Comparator): 10 obese, non-diabetic candidates will ingest SATIOSTAT as meal replacement at lunch and as first course at dinner over a period of 6 weeks. The SATIOSTAT granulates consists of hydrocolloids (fibers) and long-chain fatty acids with powder.
  Interventions: Dietary Supplement: SATIOSTAT

INTERVENTIONS:
Dietary Supplement: Control — Control granulates (maize starch and long-chain fatty acids) with powder
  Other Names: The energy content of one single bottle control is also 138kcal and contains 7.6g fat, 11.1g carbohydrates and 3.9g protein.
  Arms: Control
Dietary Supplement: SATIOSTAT — SATIOSTAT granulates (hydrocolloids (fibers) and long-chain fatty acids) with powder
  Other Names: The energy content of one single bottle SATIOSTAT is 138kcal and contains 10.5g fat, 6.4g carbohydrates and 3.9g protein.
  Arms: SATIOSTAT

SUMMARY:
SATIOSTAT is a composition comprising a specific dietary fibre component (a mixture of hydrocolloids with excellent safety profiles and a long history of use in humans) and a lipid component (long-chain fatty acids). The goal of this combination is to achieve long-acting delivery of long-chain fatty acids to the intestinal lining, triggering the sustained release of satiety-signals from intestinal cells, and consequently reducing appetite and lowering food intake in humans.

Over a period of 6 weeks, volunteers will ingest SATIOSTAT as meal replacement at lunch and as first course at dinner. Once before and after these 6 weeks the investigators will carry out an oral glucose challenge, measure satiation hormones and examine faeces (gut microbiota). Volunteers will fill in a food diary and a questionnaire for gastrointestinal symptoms and quality of life. The whole study will take approximately 8-10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Obese volunteers (BMI > 30kg/m2)
* Otherwise healthy
* Informed Consent as documented by signature (Appendix Informed Consent Form)

Exclusion Criteria:

* Food allergies, food intolerance
* Evidence of relevant cardiovascular, pulmonary, renal, hepatic, pancreatic, gastrointestinal, metabolic, endocrinological, neurological, psychiatric or other diseases at screening
* Chronic or clinically relevant acute infections
* Clinically relevant abnormalities in chemical, haematological or any other laboratory parameters
* Participation in drug trials within 2 months before start of the study
* Neurological or psychiatric disease or drug or alcohol abuse, which would interfere with the subjects proper completion of the protocol assignment
* Pregnancy: although no contraindication pregnancy might influence metabolic state. Women who are pregnant or have the intention to become pregnant during the course of the study are excluded. In female participants of childbearing age not using safe contraception (oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices) a urine pregnancy test is carried out upon screening.
* Antibiotic therapy within the last 3 months before inclusion
* Substance abuse, alcohol abuse
* Inability to follow procedures due to psychological disorders, dementia or insufficient
* Knowledge of project language (German).
* Participation in another study with investigational drug within the 30 days preceding and during the present study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Effect of chronic SATIOSTAT intake on total body weight | change from baseline to 6 weeks after SATIOSTAT intake

SECONDARY OUTCOMES:
Effect of chronic SATIOSTAT intake on glucose tolerance measured by oral glucose tolerance test | change from baseline to 6 weeks after SATIOSTAT intake
  measured with oral glucose tolerance test
Effect of chronic SATIOSTAT intake on human gut microbiota composition measured by metagenomic shotgun sequencing | change from baseline to 6 weeks after SATIOSTAT intake
  measured with metagenomic shotgun sequencing
Effect of chronic SATIOSTAT intake on gut microbial-related metabolites in feces | change from baseline to 6 weeks after SATIOSTAT intake
  Metabolomic analysis of the bacterial metabolites present in the feces by combining nuclear magnetic resonance (1H-NMR) and mass spectrometry
Effect of chronic SATIOSTAT intake on gastrointestinal symptoms assessed by questionnaire | change from baseline to 6 weeks after SATIOSTAT intake
  Assessment by use of the Gastrointestinal Symptoms Rating Scale (Svedlund et al)
Effect of chronic SATIOSTAT intake on quality of life assessed by questionnaire | change from baseline to 6 weeks after SATIOSTAT intake
  Assessment by use of the short form (SF)-36 questionnaire
Effect of chronic SATIOSTAT intake on plasma Glucagon-like Peptide (GLP-1) concentrations measured by ELISA | change from baseline to 6 weeks after SATIOSTAT intake
  measured by commercially available ELISA (enzyme-linked immunosorbent assay )-kits
Effect of chronic SATIOSTAT intake on subjective feelings of hunger and satiety measured by visual analogue scale | change from baseline to 6 weeks after SATIOSTAT intake
  measured by using visual analogue scales

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Study Chair — St. Claraspital klinische Forschungsabteilung
Locations (1):
- St Claraspital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided